CLINICAL TRIAL: NCT05176743
Title: Food Insecurity in Oncology (FIOnc)
Brief Title: Food Insecurity in Oncology
Acronym: FIOnc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: University of New Mexico Cancer Center (Other); Wake Forest University Health Sciences (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: INST UNM 2104; 5UG1CA189824-07 (NIH)
Record Dates: First submitted 2021-08-26; First posted 2022-01-04 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2021-12

CONDITIONS: Food Insecurity; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a randomized pilot trial. Eligible individuals will be identified from breast and gynecologic clinics in the New Mexico Cancer Care Alliance. Participants will be screened for food insecurity and asked to complete a baseline survey. Participants will then be randomized to either Usual Care or to the UCT intervention. All participants will complete a 3-month follow-up, survey and a qualitative exit interview.
Masking Description: No blinding will be used in this pilot trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Other): * Referral to services
  * Nutrition pamphlets
  * One-time payment of $300 paid 4 months after baseline
  Interventions: Behavioral: Unconditional Cash Transfer (UCT)
- Unconditional Cash Transfer Intervention (Experimental): * Three monthly payments of $100
  * Referral to services
  * Nutrition pamphlets
  Interventions: Behavioral: Unconditional Cash Transfer (UCT)

INTERVENTIONS:
Behavioral: Unconditional Cash Transfer (UCT) — The UCT consists of three $100 VISA merchandise cards provided monthly via mail to participants randomized to the intervention arm. Merchandise cards can be used anywhere that VISA is accepted. Participants in the UCT arm will also receive Usual Care, including referral to the patient support services team and nutritional pamphlets.

SUMMARY:
This trial will examine the feasibility and preliminary effectiveness of providing unconditional cash transfers to food insecure female breast and gynecologic cancer patients.

Approximately one-third of cancer survivors report food insecurity, characterized by limited access to adequate food for active, healthy living because of a lack of money and other resources. Unconditional cash transfers offer direct monetary assistance that can be used to meet immediate food or other financial needs and may positively impact health care resource utilization and health-related quality of life.

DETAILED DESCRIPTION:
In this delayed intervention trial, 44 female breast and gynecologic cancer patients experiencing food insecurity will be randomized in a 1:1 ratio to receive unconditional cash transfers (UCT) for 3 months or an equivalent one-time UCT at the end of the study.

Quantitative surveys will be administered at baseline and after 3-months. Survey measures will include questions about health care resource utilization, health-related quality of life, food security, hospitalization use, emergency department use, and mental health. The main objective for this pilot trial is to assess feasibility. The investigators will measure whether the investigators can: recruit 44 food insecure participants meeting the eligibility criteria over a 3-month recruitment window and describe the barriers and facilitators of the recruitment process. The investigators will also monitor retention and survey completion. At the end of the 3 month follow-up period, all participants will complete a semi-structured exit interview.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of female breast (ICD-10 C50), ovarian (ICD-10 C56), endometrial (ICD-10 C54), cervical (ICD-10 C53), vulvar cancer (ICD-10 C51)
* Diagnosed within 24-months of identification
* Stage I-III
* Completed initial course of cancer directed therapy (surgery, radiation, chemotherapy).
* Age ≥18
* Able to speak English or Spanish
* Food insecure

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Determine the percentage of referred patients who are eligible to enroll in the study and choose to do so | 3 months
Determine the percentage of patients who complete both the baseline and 3 month follow-up survey | 3 months
Determine the number of participants who complete the surveys | 3 months

SECONDARY OUTCOMES:
Assess healthcare resource utilization using the PhenX-Access to Health Services toolkit | 3 months
Healthcare costs | 3 months
Assess health-related quality of life using the PROMIS Global Health 10 item questionnaire | 3 months
  Nine of the Global Health PROMIS measures items are scored on a Likert scale, with 1 representing the worst health situation and 5 representing the best health situation. Pain is scored from 0 to 10 with 0 indicating no pain and 10 representing the worst pain ever experienced. Two sub-scores can also be derived from the 10 item questionnaire to assess physical and mental health separately. Raw scores must be converted to a standardized T-score for interpretation. A higher PROMIS T-score indicates a person whose health is better than the average respondent.
Assess the number of participants who are food insecure using the Hunger VitalSign food insecurity screening tool | 3 months
Determine the number of patients who use the Emergency Department during the 3 month follow-up period as well as how many visits they have | 3 months
Determine the number of patients who report being hospitalized during the 3 month follow-up period as well as the number of times they are hospitalized | 3 months
Assess number of participants experiencing depression using the Patient Health Questionnaire (PHQ-9) screener tool | 3 months
Assess participants perceived self-efficacy using the PROMIS Self-Efficacy for Managing Medications and Treatments 4a questionnaire | 3 months
  The 4 questions that comprise this measure are measured on a Likert scale with 1 representing that the respondent is "not at all confident" completing the described task and 5 representing that the respondent is "very confident" completing the task. Raw scores range from 4-20, but T-score conversions are needed for interpretation. A higher PROMIS T-score indicates a person whose health is better than the average respondent.
Assess incidence of participant stress using the Perceived Stress Scale (PSS-10) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean A McDougall, PhD, MPH, Principal Investigator — University of New Mexico, Internal Medicine/Epidemiology, Biostatistics & Preventive Medicine
Locations (1):
- University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No